CLINICAL TRIAL: NCT06643819
Title: A Randomized, Double-blind, Active-controlled, Multi-center, Therapeutic Confirmatory, Phase 3 Trial to Evaluate the Efficacy and Safety of CKD-202A
Brief Title: Phase 3 Trial to Evaluate the Efficacy and Safety of CKD-202A
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A119_01HTN2312
Record Dates: First submitted 2024-10-14; First posted 2024-10-16 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Valsartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test Group1 (Experimental)
  Interventions: Drug: Sacubitril∙Valsartan(dose maintenance)
- Test Group2 (Experimental)
  Interventions: Drug: Sacubitril∙Valsartan(dose increasing)
- CONTROL (Active Comparator)
  Interventions: Drug: Valsartan

INTERVENTIONS:
Drug: Sacubitril∙Valsartan(dose maintenance) — During the 4 weeks of Placebo Run-in Period(Single blind), all participants are treated 1 placebo of CKD-202A(Sacubitril∙Valsartan) 100mg and 1 placebo of D763(Valsartan 80 mg) each, total of 2 oral doses once a day.
  After Placebo Run-in Period, During the 4 weeks out of 10 weeks of Treatment Period(Double blind), All TEST1 pariticipants are treated 1 CKD-202A (Sacubitril∙Valsartan) 100 mg and 1 placebo of D763(Valsartan 80 mg) each, total of 2 oral doses once a day.
  After 4 weeks of Treatment Period, During the 6 weeks out of 10 weeks of Treatment Period(Double blind), All TEST1 pariticipants are treateed 1 CKD-202A (Sacubitril∙Valsartan) 100 mg, 1 placebo of CKD-202A(Sacubitril∙Valsartan) 200mg, 1 placebo of D764(Valsartan 160 mg) each, and a total of 3 oral doses once a day.
  Arms: Test Group1
Drug: Sacubitril∙Valsartan(dose increasing) — During the 4 weeks of Placebo Run-in Period(Single blind), all participants are treated 1 placebo of CKD-202A(Sacubitril∙Valsartan) 100mg and 1 placebo of D763(Valsartan 80 mg) each, total of 2 oral doses once a day.
  After Placebo Run-in Period, During the 4 weeks out of 10 weeks of Treatment Period(Double blind), All TEST2 pariticipants are treated 1 CKD-202A (Sacubitril∙Valsartan) 100 mg and 1 placebo of D763(Valsartan 80 mg) each, total of 2 oral doses once a day.
  After 4 weeks of Treatment Period, During the 6 weeks out of 10 weeks of Treatment Period(Double blind), All TEST1 pariticipants are treateed 1 placebo of CKD-202A (Sacubitril∙Valsartan) 100 mg, 1 CKD-202A(Sacubitril∙Valsartan) 200mg, 1 placebo of D764(Valsartan 160 mg) each, and a total of 3 oral doses once a day.
  Arms: Test Group2
Drug: Valsartan — During the 4 weeks of Placebo Run-in Period(Single blind), all participants are treated 1 placebo of CKD-202A(Sacubitril∙Valsartan) 100mg and 1 placebo of D763(Valsartan 80 mg) each, total of 2 oral doses once a day. After Placebo Run-in Period, During the 4 weeks out of 10 weeks of Treatment Period(Double blind), All TEST2 pariticipants are treated 1 placebo of CKD-202A (Sacubitril∙Valsartan) 100 mg and 1 D763(Valsartan 80 mg) each, total of 2 oral doses once a day. After 4 weeks of Treatment Period, During the 6 weeks out of 10 weeks of Treatment Period(Double blind), All TEST1 pariticipants are treateed 1 placebo of CKD-202A (Sacubitril∙Valsartan) 100 mg, 1 placebo of CKD-202A(Sacubitril∙Valsartan) 200mg, 1 D764(Valsartan 160 mg) each, and a total of 3 oral doses once a day.
  Arms: CONTROL

SUMMARY:
Phase 3 Trial to Evaluate the Efficacy and Safety of CKD-202A(Sacubitril∙Valsartan)

ELIGIBILITY:
Inclusion Criteria:

* Participants who are 19 years old or older.
* Participants who have voluntarily decided to participate in this clinical trial and signed ICF.

Exclusion Criteria:

* Participants with a history of secondary hypertension or suspected secondary hypertension.
* Participants with a orthostatic hypotension.
* Participants who require combination administration of antihypertensive drugs other than clinical trial drugs during the clinical trial participation period.
* Participants with type 1 diabetes or poorly controlled diabetes.
* Participants who treated other clinical trial drugs within 4 weeks of screening visit.
* Participants with a history of drug or alcohol abuse or suspected patient within 24 weeks as of the time of screening
* Pregnant women, lactating women, or Subjects who do not agree to use appropriate contraception during the clinical trial period and for two weeks after the end of administration of the last clinical trial drug
* Participants who are unable to participate in this clinical trial at the discretion of the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2024-10-14 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
change from baseline in MASBP(Mean Ambulatory Systolic Blood Pressure) | 10 weeks after baseline
  The purpose of Clinical Trial is confirmation that test group 2 (Sacubitril∙Valsartan 200mg) is superior to control group (Valsartan 160mg)

CONTACTS AND LOCATIONS:
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, South Korea

IPD SHARING:
Plan to Share IPD: No